CLINICAL TRIAL: NCT05030662
Title: National Taipei University of Nursing and Health Sciences
Brief Title: Walking Stick Exercise in Patients Underwent Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Responsible Party: Principal Investigator, Yu Hua Chou, Principal Investigator, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YChou
Record Dates: First submitted 2021-08-14; First posted 2021-09-01 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Arthroplasty; Replacement; Knee Osteoarthritis
Keywords: total knee arthroplasty; Walking stick exercise
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Masking Description: Sigle,were not involved in the study assessments beyond recording the timed-get-up-and-go test before and after the treatment intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental:Walking stick exercise (Experimental): The experimental:Walking stick exercise
  1. Education of walking stick exercise by research nurses twice before discharge (on the day before surgery and before discharge)
  2. The video clip of "walking stick exercise" is available to the patients.
  3. The research nurses encourage our patients to keep rehabilitation by phone calls once a week after discharge.
  Interventions: Other: Walking stick exercise
- Control group: conventional physical therapy. (No Intervention): 1. Perform bed mobility and transfers with the least amount of assistance while maintaining appropriate weight bearing (WB) precautions.
  2. Ambulate with an assistive device for 25-100 feet and ascend/descend stairs to allow for independence with household activities while maintaining appropriate WB.
  3. Verbalize understanding of post-operative activity recommendations/precautions including use of proper positioning of the lower extremity, range of motion and strengthening exercises.

INTERVENTIONS:
Other: Walking stick exercise — 1. Education of walking stick exercise by research nurses twice before discharge (on the day before surgery and before discharge)
  2. The video clip of "walking stick exercise" is available to the patients.
  3. The research nurses encourage our patients to keep rehabilitation by phone calls once a week after discharge.
  Arms: Experimental:Walking stick exercise

SUMMARY:
The purpose of this study is to examine whether the effect of "hiking poles exercise" on lower extremity muscular strength, knee range of motion, and quality of life in elderly patients underwent total knee arthroplasty

DETAILED DESCRIPTION:
This is a longitudinal-experimental study. The data collection and analysis are in a single-blind manner. The study will be undertaken in the Department Orthopaedics of En Chu Kong hospital (approximate 500-bed regional teaching hospital). All patients who meet the inclusion criteria are admitted for primary total knee arthroplasty and assigned to control group or intervention group randomly. The 44 patients in the control group received routine guidance of " Rehabilitation and precautions for artificial knee replacement ". In addition to the routine guidance, the 44 patients in the intervention group received educations of " hiking poles exercise " on the day before surgery and before discharge, as well as a follow-up call at least once a week after discharge.

ELIGIBILITY:
Minimum Age: 60 years Maximum Age: 85years Gender-Based: All Accepts Healthy Volunteers:No

Criteria:

Inclusion Criteria:

* Age between 60 and 85 years
* Informed consent
* Receipt of elective unilateral primary knee arthroplasty surgery.

Exclusion Criteria:

* Non-degenerative arthritis, including rheumatoid arthritis, or traumatic arthritis
* Patients receiving rehabilitation simultaneously
* Patients with other musculoskeletal or neurological problems, including fractures, Parkinsonism, cerebrovascular events, or patients with multiple comorbidities
* Cancer patients receive chemotherapy
* Patients with the peri-operative complication that has an adverse effect on outcomes,for example: intra-operative fractures, thromboembolism, peri-operative infections, or phlebitis

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Total knee arthroplasty of Quality of life | for three months
  I hope the Walking stick exercise can to improving the total knee arthroplasty quality of life of patients. I use Knee injury and Osteoarthritis Outcome Score (KOOS). There are 5 territories analyzed in the knee injury and osteoarthritis outcome score (KOOS) calculator and a knee-related QOL, Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopedic scales and generic measures. Scores between 0 and 100 represent the percentage of the total possible score achieved. Furthermore, I will follow up to study on the day before surgery at 1, 6, and 12 weeks post-surgery.

SECONDARY OUTCOMES:
lower limb muscle power | for three months
  I hope the Walking stick exercise can to improving the total knee arthroplasty lower limb muscle power. I use include 30-second chair stand test. Furthermore, I will follow up to study on the day before surgery at 1, 6, and 12 weeks post-surgery.
knee range of motion | for three months
  I hope the Walking stick exercise can to improving the total knee arthroplasty lower limb muscle power. I use include 30-second chair stand test. Furthermore, I will follow up to study on the day before surgery at 1, 6, and 12 weeks post-surgery.

OTHER OUTCOMES:
participant characteristics | on the day before surgery
  age, sex, body mass index, job occupation, marriage,Primary caregiver, Exercise habits, BMI % , and education

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hua Chou, Principal Investigator — none,specify Unaffiliated
Locations (1):
- TAIWAN, New Taipei City, Taiwan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-08-01): https://cdn.clinicaltrials.gov/large-docs/62/NCT05030662/Prot_ICF_000.pdf